CLINICAL TRIAL: NCT00894816
Title: Effects of Feeding Lactobacillus F19 to Infants During Weaning on Allergies, Immune Programming, Gut Microbiota, Overweight and Oral Health
Brief Title: Probiotics in Prevention of Allergies, Obesity and Caries
Acronym: ELEFANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Karolinska Institutet (Other); University of Helsinki (Other); The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); Medical Research Council (Other Government); Ekhagastiftelsen (Other); The county of Västerbotten (Unknown); Oskar Foundation (Other)
Responsible Party: Principal Investigator, Christina West, Dr, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ELEFANT
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Eczema; Allergy; Asthma; Obesity; Dental Caries
Keywords: Prevention; Probiotics; Eczema; Allergy; Asthma; Obesity; Caries; Gut microbiota
MeSH Terms: conditions — Eczema; Hypersensitivity; Asthma; Obesity; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Infant cereals with the addition of Lactobacillus paracasei subsp. paracasei strain F19 (LF19) 10E8 CFU per serving
  Interventions: Dietary Supplement: Lactobacillus F19
- 2 (Placebo Comparator): Placebo (infant cereals without any additions)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus F19 — Infant cereals with the addition of Lactobacillus paracasei subsp. paracasei strain F19 (LF19)10E8 CFU per serving
  Arms: 1
Dietary Supplement: Placebo — Infant cereals without any addition
  Arms: 2

SUMMARY:
During the period of 2000-2003, 179 healthy, term infants with no previous signs of allergic disease were recruited and randomized to daily intake of cereals with or without the addition of Lactobacillus paracasei subspecies paracasei strain F19 (LF19) from 4-13 months of age. The effects of LF19 on gut microbial composition, infections, allergies, immunological development, growth and blood lipids were monitored. Of 179 included infants, 171 completed the study. The study product was well tolerated with no observed side effects. Compliance was excellent.

In a follow-up study, the aim is to investigate the long-term effects of feeding LF19 during weaning on allergies, immune programming, overweight, gut microbial composition and oral health in 8-year old children.

The investigators' primary outcome will be to determine whether daily intake of LF19 during weaning results in less eczema at 8 years of age, and if the preventive effect encompasses also respiratory allergies and immunoglobulin E (IgE) - sensitization. The long term effects on gut microbial composition, overweight and metabolic markers will be investigated. Furthermore, the possible preventive effects of LF19 on caries will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants born at term (gestational age 37-42 weeks)
* Birth weight > 2500 g
* Vaginally delivered
* No atopic manifestation
* A normal diet for age
* No medication that could have affected the intestinal microbiota

Ages: 4 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2000-08; Primary Completion 2011-09 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Eczema | 8 years of age
  Eczema including related allergic manifestations

SECONDARY OUTCOMES:
Respiratory allergies | 8 years of age
  Allergic rhinitis and asthma
Sensitization | 8 years of age
  Assessed by skin prick test and specific IgE tests
Overweight/obesity | 8 years of age
  Assessed by BMI and DEXA-scan
Gut microbial composition | 8 years of age
  Assessed by Molecular biology techniques
Caries | 8 years of age
  Clinical evaluation and x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Christina E West, MD, PhD, Principal Investigator — Clinical Sciences, Pediatrics, Umeå University, SE-901 87 Umeå, Sweden; Olle Hernell, Professor, Study Chair — Clinical Sciences, Pediatrics, Umeå University, SE-901 87 Umeå, Sweden
Locations (1):
- Umeå University, Umeå, Sweden

REFERENCES:
- [Background] Karlsson Videhult F, Ohlund I, Stenlund H, Hernell O, West CE. Probiotics during weaning: a follow-up study on effects on body composition and metabolic markers at school age. Eur J Nutr. 2015 Apr;54(3):355-63. doi: 10.1007/s00394-014-0715-y. Epub 2014 May 17. PMID 24830782
- [Result] West CE, Gothefors L, Granstrom M, Kayhty H, Hammarstrom ML, Hernell O. Effects of feeding probiotics during weaning on infections and antibody responses to diphtheria, tetanus and Hib vaccines. Pediatr Allergy Immunol. 2008 Feb;19(1):53-60. doi: 10.1111/j.1399-3038.2007.00583.x. Epub 2007 Dec 11. PMID 18086218
- [Result] West CE, Hammarstrom ML, Hernell O. Probiotics during weaning reduce the incidence of eczema. Pediatr Allergy Immunol. 2009 Aug;20(5):430-7. doi: 10.1111/j.1399-3038.2009.00745.x. Epub 2009 Mar 9. PMID 19298231
- [Result] West CE, Hernell O, Andersson Y, Sjostedt M, Hammarstrom ML. Probiotic effects on T-cell maturation in infants during weaning. Clin Exp Allergy. 2012 Apr;42(4):540-9. doi: 10.1111/j.1365-2222.2011.03941.x. PMID 22417212
- [Result] West CE, Hammarstrom ML, Hernell O. Probiotics in primary prevention of allergic disease--follow-up at 8-9 years of age. Allergy. 2013 Aug;68(8):1015-20. doi: 10.1111/all.12191. Epub 2013 Jul 30. PMID 23895631
- [Result] Hasslof P, West CE, Videhult FK, Brandelius C, Stecksen-Blicks C. Early intervention with probiotic Lactobacillus paracasei F19 has no long-term effect on caries experience. Caries Res. 2013;47(6):559-65. doi: 10.1159/000350524. Epub 2013 Jul 4. PMID 23838478